CLINICAL TRIAL: NCT01017887
Title: SurgiQuest AirSeal CO2 Gas Quality
Brief Title: Intraperitoneal Carbon Dioxide Concentration Measurement During Standard Laparoscopy With a New Airseal Access Port
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit any subjects
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, David Earle, MD, Baystate Medical Center
Other Study IDs: IRB09-107
Record Dates: First submitted 2009-08-04; First posted 2009-11-23 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Laparoscopic Carbon Dioxide Measurement
Keywords: laparoscopy; airseal; carbon dioxide; insufflation; pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Airseal port for laparoscopic surgery: Airseal access port for laparoscopic surgery with standard ports.
  Interventions: Device: Airseal access port for laparoscopic surgery; Device: Standard Laparoscopy ports
- Standard Laparoscopy ports: Uses standard laparoscopy ports.
  Interventions: Device: Standard Laparoscopy ports

INTERVENTIONS:
Device: Airseal access port for laparoscopic surgery — The investigators will utilize this access port that is already approved by the FDA for it's intended use in laparoscopic surgery. The investigators are simply measuring the percentage of carbon dioxide in the peritoneal cavity.
  Groups: Airseal port for laparoscopic surgery
Device: Standard Laparoscopy ports — Prospective monitoring of CO2 levels during laparoscopic surgery with standard access ports.

SUMMARY:
The new AirSeal access port for laparoscopic surgery does not use a mechanical valve on the port to maintain gas in the peritoneal cavity. It uses an invisible barrier created by high flow gas jets within the port. The percentage of carbon dioxide, the standard gas used for laparoscopy, during laparoscopic surgery has not been previously measured, but is probably high. The investigators aim to measure the percentage of intraperitoneal carbon dioxide with standard ports and the AirSeal port during a variety of conditions during laparoscopic procedures including suturing and suctioning. The study period will commence at the start of the operation, and be completed upon discharge from the hospital or postoperative day 5, whichever is shorter. All devices are approved for use in humans by the FDA, and are being used for their intended purpose.

DETAILED DESCRIPTION:
The SurgiQuest AirSeal system is approved by the Food and Drug Administration (FDA) as access port for laparoscopic surgery that utilizes an invisible air curtain rather than a mechanical barrier to maintain pneumoperitoneum. In addition to the cannula, there is special filtration tubing and an air pump that act in concert with an existing CO2 insufflator. The system has been approved for use and purchase at Baystate Medical Center by the value analysis committee. Despite FDA approval and extensive laboratory testing, there is still no human data regarding intraperitoneal CO2 levels under a variety of conditions one would normally experience during a laparoscopic operation. The specific aim of this study is to measure these levels during laparoscopic cases in humans. We hypothesize that there will be no more than minimal alteration of intraperitoneal CO2 levels when using the AirSeal system when compared to the standard laparoscopic system. The follow-up to this is examining evidence of extraperitoneal gas extravasation. This will occur as part of routine post-operative care, but we will be collecting data, that will be de-identified in the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a laparoscopic operation

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing a laparoscopic operation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
percent of intraperitoneal carbon dioxide during surgery | intraoperative - starts at beginning of the operation and ends at the completion of the operation
  intraperitoneal carbon dioxide measurements intraoperatively

SECONDARY OUTCOMES:
subcutaneous emphysema | during the patients hospital stay, or the first 5 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: David Earle, MD, Principal Investigator — Baystate Medical Center